CLINICAL TRIAL: NCT06276140
Title: Preoperative Evaluation and Impact of Iron Deficiency Anaemia on the Incidence of Perioperative Complications and Quality of Recovery After Radical Colorectal Cancer Surgery
Brief Title: Iron-deficiency Anaemia and Its Impact on Recovery After Colorectal Cancer Surgery
Acronym: ID-COLO
Status: Enrolling by invitation | Type: Observational
Sponsor: Oncology Institute of Vojvodina (Other Government)
Collaborators: University of Bern (Other)
Responsible Party: Principal Investigator, Nora Mihalek, Dr., Oncology Institute of Vojvodina
Other Study IDs: 4/23/2-4661/2-9
Record Dates: First submitted 2024-02-18; First posted 2024-02-23 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Iron Deficiencies; Iron Deficiency Anaemia; Postoperative Complications; Colorectal Cancer
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency; Postoperative Complications; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for laboratory analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Iron deficiency anaemia: Defined as: decreased serum iron concentration and TSAT, increased TIBC, UIBC, as well as decreased haemoglobin concentration (HGB)
  Interventions: Diagnostic Test: Laboratory analyses for the detection of iron deficiency anaemia
- Iron deficiency in the latent phase: Defined as: decreased serum iron concentration and TSAT, increased TIBC, UIBC, as well as normal HGB
  Interventions: Diagnostic Test: Laboratory analyses for the detection of iron deficiency anaemia
- Control group: Defined as: normal serum iron concentration, TSAT, TIBC, UIBC and HGB
  Interventions: Diagnostic Test: Laboratory analyses for the detection of iron deficiency anaemia

INTERVENTIONS:
Diagnostic Test: Laboratory analyses for the detection of iron deficiency anaemia — Erythrocyte indices based on the preoperative complete blood count results will be calculated for each patient one day prior to surgical treatment.
  Overall morbidity of each patient during hospital stay will be scored using the Comprehensive Complication Index (CCI). Intraoperative complications will be graded according to the ClassIntra classification of intraoperative adverse events. The quality of postoperative recovery of each observed patient will be scored on the first, second and fifth postoperative day, using the 15-item quality of recovery scale (QoR-15).
  Data about red blood cell transfusion rate, all-cause infection rate, number of days when antibiotics were administered and the number of different antibiotics administered during hospital-stay will be collected.

SUMMARY:
The aim of this prospective, observational cohort study is to assess the impact of iron deficiency anaemia on the incidence of perioperative complications and the quality of recovery after surgery in patients undergoing colorectal cancer surgery. The main questions the study aims to answer are:

* whether the presence of preoperative iron deficiency anaemia leads to a poorer quality of postoperative recovery in patients undergoing colorectal cancer surgery
* whether different combinations of complete blood count parameters (red blood cell indices) could be suitable diagnostic tools for the detection of iron deficiency in the latent stage (without laboratory-confirmed anaemia) in colorectal cancer patients.

Blood samples for laboratory analyses will be collected from each study patient admitted to the surgical ward one day prior to elective surgery and on the first postoperative day during the stay in the intensive care unit. The pre-operative laboratory analyses include a complete blood count and serum iron status parameters (iron concentration, ferritin concentration, TIBC, UIBC and TSAT). Laboratory parameters analysed on the first postoperative day include complete blood count, serum concentration of electrolytes (Na, K, Ca, Cl, Mg), serum concentration of urea and creatinine, parameters of haemostasis (aPTT, PT, INR), serum concentration of C-reactive protein and procalcitonin.

Data about overall morbidity, intraoperative complications, quality of postoperative recovery, red blood cell transfusion rate, all-cause infection rate, antibiotic usage, as well as length of hospital stay will be collected.

The researchers will compare the group of patients with iron deficiency anaemia, the group of patients with iron deficiency in the latent stage and the control group to determine whether patients with iron deficiency have a higher incidence of perioperative complications and impaired recovery after surgery. The researchers will investigate whether iron deficiency can be detected at an early stage, when anaemia is not yet present, by calculating various red blood cell indices.

DETAILED DESCRIPTION:
The following erythrocyte indices based on the preoperative complete blood count results will be calculated for each patient one day prior to surgical treatment:

* Mentzer index: MCV / RBC
* Green and King index: MCV2 x RDW / (100 x HGB)
* RDW index: MCV x RDW / RBC
* Shine and Lal index: MCV2 x MCH / 100
* England and Fraser index: MCV - RBC - (5 x HGB) - 3.4
* Srivastava index: MCH / RBC
* Ricerca index: RDW / RBC
* Ehsani index: MCV - (10 x RBC)
* Sirdah index: MCV - RBC - (3 x HGB)
* Sehgal index: MCV2 / RBC

The Ganzoni equation for calculating total iron deficit will be calculated for each patient one day prior to surgical treatment, using the following formula:

total iron deficit [mg] = body weight [kg] x (target hemoglobin [g/L] - actual hemoglobin [g/L]) x 2.4 + iron depot [mg]

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (˃ 18 years of age)
* ASA III clinical status
* Patients undergoing radical surgical treatment of colorectal cancer
* Signed written informed consent

Exclusion Criteria:

* Patients undergoing palliative surgical treatment of colorectal cancer
* Anaemic patients without iron deficiency, defined as: normal serum iron concentration, TSAT, TIBC, UIBC, and decreased HGB, HCT and RBC
* Presence of other type of anaemia than iron deficiency anaemia (e.g. alpha- or beta-thalassemia, sickle-cell anaemia, etc.)
* History of red blood cell transfusion in the period of 120 days prior to hospital-admission
* Stage III, IV, or V of chronic kidney disease (creatinine clearance < 60 mL/min)
* Significant intraoperative bleeding, which requires transfusion of red blood cell products, calculated using the Gross-formula:

allowable blood loss [mL] = (estimated blood volume [mL] x (initial HGB [g/L] - HGB level when transfusion is required [g/L])) / average of initial HGB and HGB level when transfusion is required [g/L] The cut-off value for HGB level when transfusion is required is set to 80 g/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing elective surgical treatment of colorectal cancer.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Overall morbidity | during hospital-stay
  score of Comprehensive Complication Index (CCI)

SECONDARY OUTCOMES:
Prevalence of absolute iron deficiency, functional iron deficiency and iron deficiency anaemia in the study population | at inclusion
  number of patients; proportion
Red blood cell transfusion rate | during hospital-stay
  number of cases; proportion
All-cause infection rate | during hospital-stay
  number of cases; proportion
Days of antibiotic use | during hospital-stay
  number of days
Number of different antibiotics administered | during hospital-stay
  number of antibiotics
Length of Intensive care unit-stay | during hospital-stay
  number of days
Length of hospital-stay | during hospital-stay
  number of days
Intraoperative complications | during anaesthesia and surgical intervention
  grade of ClassIntra classification of intraoperative adverse events
Quality of postoperative recovery | on the first, second and fifth postoperative day
  score achieved on QoR-15 scale
Reoperation | during hospital-stay
  number of cases; proportion
Estimated total iron-deficit | one day prior to surgery
  in mg, using the Ganzoni equation
Serum ferritin level | one day prior to surgery
  in ng/mL
Values of different erythrocyte indices | one day prior to surgery
  calculated based on the complete blood count parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Institute of Vojvodina, Kamenitz, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slankamenac K, Graf R, Barkun J, Puhan MA, Clavien PA. The comprehensive complication index: a novel continuous scale to measure surgical morbidity. Ann Surg. 2013 Jul;258(1):1-7. doi: 10.1097/SLA.0b013e318296c732. PMID 23728278
- [Background] Krielen P, Gawria L, Stommel MWJ, Dell-Kuster S, Rosenthal R, Ten Broek RPG, van Goor H. Inter-Rater Agreement of the Classification of Intraoperative Adverse Events (ClassIntra) in Abdominal Surgery. Ann Surg. 2023 Feb 1;277(2):e273-e279. doi: 10.1097/SLA.0000000000005024. Epub 2023 Jan 10. PMID 34171869
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Al-Naseem A, Sallam A, Choudhury S, Thachil J. Iron deficiency without anaemia: a diagnosis that matters. Clin Med (Lond). 2021 Mar;21(2):107-113. doi: 10.7861/clinmed.2020-0582. PMID 33762368
- [Background] Cappellini MD, Musallam KM, Taher AT. Iron deficiency anaemia revisited. J Intern Med. 2020 Feb;287(2):153-170. doi: 10.1111/joim.13004. Epub 2019 Nov 12. PMID 31665543